CLINICAL TRIAL: NCT01607866
Title: Quadrant Parotidectomy Versus Superficial Parotidectomy for Treatment of Pleomorphic Adenoma
Brief Title: Quadrant Versus Superficial Parotidectomy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment of eligible patients for randomization.
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Associate Professor of Surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R/89
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Pleomorphic Adenoma of the Parotid Gland

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadrant parotidectomy (Experimental): Patients in this arm will receive excision of the parotid gland quadrant harboring the tumor
  Interventions: Procedure: Quadrant parotidectomy
- Superficial parotidectomy (Active Comparator): Patients in this group will receive superficial parotidectomy
  Interventions: Procedure: Superficial parotidectomy

INTERVENTIONS:
Procedure: Quadrant parotidectomy — Excision of one quadrant of the parotid gland which is comparable to half of the superficial lobe of the gland
  Arms: Quadrant parotidectomy
Procedure: Superficial parotidectomy — Excision of the whole superficial lobe of the parotid gland
  Arms: Superficial parotidectomy

SUMMARY:
The most common benign tumor of the parotid gland is the so called pleomorphic adenoma. Although benign, this tumor may recur after surgical removal due to tumor cells left behind during the surgical operation. Thus, pleomorphic adenomas have been treated with wide resection similar to malignant tumors. This extensive surgery often leads to injury to the motor nerves responsible for facial expression and eye protection. The investigators propose less extensive surgery which should be thorough enough to prevent tumor recurrence while keeping the facial nerve out of risk.

DETAILED DESCRIPTION:
Pleomorphic adenoma is notorious of its propensity to local recurrence due to the microscopic extracapsular extension of the tumor. Superficial parotidectomy (SP) is the standard treatment. Extracapsular dissection (ED) has been proposed to minimize the risk of facial nerve palsy. However, the oncologic safety of ED is controversial in the literature. We propose quadrant parotidectomy (QP) which is less radical than SP and less conservative than ED. QP entails dissection overlying one primary division of the facial nerve leaving the other division undisturbed while the resection safety margin is still generous.

Surgery for pleomorphic adenoma is a compromise between radicality and facial nerve morbidity. Risk of local recurrence is imprecisely described in the literature and is universally regarded as infrequent and remote. Many studies did not report recurrent cases. Thus, Facial nerve injury is the main concern of parotid surgeons and is considered the primary end point of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pleomorphic adenoma of the parotid gland with Cytology- proven diagnosis

Exclusion Criteria:

* Collagen diseases
* Previous parotid surgery
* Previous facial nerve palsy
* Neuromuscular diseases affecting the face
* Patient refusal

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with permanent facial nerve palsy | measured six months after the date of surgery
  using clinical neurological examination

SECONDARY OUTCOMES:
Number of participants with temporary facial nerve palsy | Measured at one day and at three months from the date of surgery.
  using clinical neurological examination
Operative time in minutes | Measured at the time of surgery
  Median and range of operative time per intervention arm will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hussein, MD, PhD, Principal Investigator — Mansoura University; Adel Denewer, MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University Cancer Center, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Uyar Y, Caglak F, Keles B, Yildirim G, Salturk Z. Extracapsular dissection versus superficial parotidectomy in pleomorphic adenomas of the parotid gland. Kulak Burun Bogaz Ihtis Derg. 2011 Mar-Apr;21(2):76-9. doi: 10.5606/kbbihtisas.2011.003. PMID 21417969
- [Background] Prichard AJ, Barton RP, Narula AA. Complications of superficial parotidectomy versus extracapsular lumpectomy in the treatment of benign parotid lesions. J R Coll Surg Edinb. 1992 Jun;37(3):155-8. PMID 1328626